CLINICAL TRIAL: NCT04456166
Title: Safety of Preoperative Carbohydrate Loading in Diabetic Patients Undergoing General Anesthesia
Brief Title: Safety of Preoperative Carbohydrate Loading in Diabetic Patients
Acronym: NoNPO
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Susie Yoon, Clinical Assistant Professor, Seoul National University Hospital
Other Study IDs: 20030471108
Record Dates: First submitted 2020-06-25; First posted 2020-07-02 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Carbohydrate Intolerance; Diabetes Mellitus Type 2
Keywords: Carbohydrate Intolerance; Diabetes Mellitus; Diabetes Mellitus, Type 2; Carbohydrate loading
MeSH Terms: conditions — Glucose-Galactose Malabsorption; Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient who received carbohydrate loading: Patients with diabetes mellitus type 2 who are planned to receive a carbohydrate beverage (400 ml (12.8% carbohydrates, 50 kcal/100 ml; Nucare NONPO Ⓡ , Daesang Wellife, Korea) before the operation and up to 2 hours before the induction of anesthesia outside this clinical study setting
  Interventions: Dietary Supplement: noNPO

INTERVENTIONS:
Dietary Supplement: noNPO — Patients with diabetes mellitus type 2 who are planned to receive a carbohydrate beverage (400 ml (12.8% carbohydrates, 50 kcal/100 ml; Nucare NONPO Ⓡ , Daesang Wellife, Korea) before the operation and up to 2 hours before the induction of anesthesia outside this clinical study setting will be asked to be enrolled into the study.
  Before induction of general anesthesia, all patients were evaluated the gastric volume under ultrasonography.

SUMMARY:
The purpose of this study is to investigate the safety of preoperative carbohydrate loading in diabetic patients undergoing general anesthesia

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery
* Type 2 diabetes mellitus on oral hypoglycemic agents
* American Society of Anesthesiologists physical status 2 or 3
* Ages 18 or more
* Approve to participate

Exclusion Criteria:

* Ambulatory surgery
* BMI >35
* History of gastric or esophagus surgery
* History of GERD, dyspepesia or
* Anticipated difficult intubation (previous III or more Cormack and Lehane's grade, Mallamgrade, Mallampati scpati scoreore III or moreIII or more, propro/retro/retrognathism, gnathism, thyromental distance<6.5cm, thyromental distance<6.5cm, limited mouth openinglimited mouth opening)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years of age who are scheduled to undergo general anesthesia are subject to preoperative carbohydrodritate loading and diagnosed with type 2 diabetes taking oral hypoglycemic agents
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-06-22 (Actual); Primary Completion 2021-05-04 (Actual); Study Completion 2021-05-04 (Actual)

PRIMARY OUTCOMES:
Incidence of gastric ultrasonography score as low risk (grade 0 or 1) | 30 minutes after intubation
  Ultrasound assessment of gastric volume by gastroscopic examination.

SECONDARY OUTCOMES:
Gastric volume | 30 minutes after intubation
Blood sugar test | 30 minutes after intubation and 30 minutes after extubation
The incidence of insulin bolus injection | during operation
The incidence of insulin bolus injection | up to 30 minutes after extubation
Satisfaction scale of patients | up to 30 minutes after extubation
The incidence of nausea and vomiting | up to 30 minutes after extubation

CONTACTS AND LOCATIONS:
Overall Officials: Susie Yoon, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Jongnogu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lee S, Sohn JY, Lee HJ, Yoon S, Bahk JH, Kim BR. Effect of pre-operative carbohydrate loading on aspiration risk evaluated with ultrasonography in type 2 diabetes patients: a prospective observational pilot study. Sci Rep. 2022 Oct 20;12(1):17521. doi: 10.1038/s41598-022-21696-1. PMID 36266449